CLINICAL TRIAL: NCT05917509
Title: A Phase IIIb, Multi-center, Non-randomized, Parallel-group, Open-label, Hybrid Type I Study Evaluating the Efficacy, Safety, Implementation Effectiveness, and Patient-reported Outcomes of Oral Dolutegravir/Lamivudine Once-daily as a First-line Regimen Followed by Participant-determined Optional Switch to Long-acting Intramuscular Cabotegravir Plus Rilpivirine Every Two Months for the Maintenance of Virologic Suppression in Antiretroviral Therapy Naive Adults Living With HIV-1
Brief Title: A Study to Evaluate the Efficacy, Safety, Participant Choice and Preference of an Oral Once-daily Regimen or a Long-acting Injectable Regimen Every Two Months for Treatment of Human Immunodeficiency Virus (HIV-1) in Adults Who Have Not Previously Taken Antiretroviral Therapy
Acronym: VOLITION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219700; 2023-503893-19-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-06-13; First posted 2023-06-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV-1; dolutegravir; lamivudine; cabotegravir; rilpivirine; Antiretroviral therapy (ART) - naïve; optional switch study; Long-acting; Fixed-dose combination; People living with HIV (PLHIV); Integrase inhibitor
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants Receiving DTG/3TC Fixed Dose Combination (FDC) (Experimental)
  Interventions: Drug: DTG/3TC
- Participants Receiving CAB + RPV LA (Experimental)
  Interventions: Drug: Cabotegravir (CAB) LA; Drug: Rilpivirine (RPV) LA

INTERVENTIONS:
Drug: DTG/3TC — DTG/3TC FDC will be administered as an oral once daily tablet.
  Other Names: Dovato
  Arms: Participants Receiving DTG/3TC Fixed Dose Combination (FDC)
Drug: Cabotegravir (CAB) LA — CAB LA will be administered as a gluteal intramuscular injection once every 2 months in combination with RPV LA.
  Other Names: Vocabria
  Arms: Participants Receiving CAB + RPV LA
Drug: Rilpivirine (RPV) LA — RPV LA will be administered as a gluteal intramuscular injection once every 2 months in combination with CAB LA.
  Other Names: Rekambys
  Arms: Participants Receiving CAB + RPV LA

SUMMARY:
This is a multicentre study carried out in participants living with human immunodeficiency virus type 1 (HIV-1) who have not previously been treated with any antiretroviral therapies. The study will investigate two 2-drug regimens for the treatment of HIV-1: a fixed-dose combination oral tablet of dolutegravir/lamivudine (DTG/3TC) and cabotegravir plus rilpivirine long-acting agents (CAB + RPV LA). All participants will initially receive DTG/3TC once daily, and once virologic suppression is attained (plasma HIV-1 <50 c/mL), participants will be offered a choice to switch to CAB + RPV LA or to continue taking oral DTG/3TC. This study will provide important data on the efficacy, safety, implementation effectiveness, and patient-reported outcomes of these two regimens in a study where participants have the option to choose between them based on individual preference. The aim of the study is to evaluate the antiviral effectiveness at 11 months after switching to CAB+RPV LA following initial virologic suppression on DTG/3TC and to provide data on how long it takes participants to suppress their viral load on DTG/3TC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with plasma HIV-1 RNA ≥1,000 c/mL at Screening.
2. Antiretroviral-naïve participants (defined as no prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection) prior to enrolment.
3. Participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
4. Participants enrolled in France must be affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study.
2. Participants with any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease; with the exception of cutaneous Kaposi's sarcoma not requiring systemic therapy, and CD4+ count <200 cells/cubic millimetre (mm^3) (neither is exclusionary).
3. Participants with history or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates study participation.
4. Participants with ongoing or clinically relevant pancreatitis.
5. Participants with Clinically significant cardiovascular disease, as defined by recent history (within the last 6 months) or current evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
6. Corrected QT (QTc) interval >450 milliseconds (msec) (or QTc >480 msec for participants with bundle branch block).
7. Participants with ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the Investigator and the Medical Monitor for inclusion of the participant prior to enrolment.
8. Participants with hereditary coagulation and platelet disorders (e.g., haemophilia or von Willebrand Disease); or current or anticipated need for chronic anti-coagulation, with the exception of the use of low-dose acetylsalicylic acid (≤325 mg).
9. Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
10. Participants with unstable liver disease as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis, or decompensated cirrhosis (e.g., ascites, encephalopathy, or variceal bleeding), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per Investigator assessment).
11. Participants with history of liver cirrhosis with or without hepatitis viral co-infection.
12. Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment.
13. Participants who, in the Investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
14. Participants with signs and symptoms which, in the opinion of the Investigator, are suggestive of active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 14 days prior to enrolment.
15. Evidence of hepatitis B virus (HBV) infection based on the results of testing at Screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), and hepatitis B surface antibody (anti-HBs) as follows:

    * Participants positive for HBsAg are excluded
    * Participants negative for HBsAg and negative for anti-HBs but positive for anti-HBc are excluded only if HBV DNA is detected [either detected below lower limit of quantification (LLOQ); detected above upper limit of quantification (ULOQ); or numerical value (i.e. between LLOQ and ULOQ)];
    * Participants negative for HBsAg but positive for anti-HBc and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
16. Participants with hepatitis C virus (HCV) co-infection at Screening are eligible only if:

    * liver enzymes meet entry criteria; and
    * HCV disease is not anticipated to require on-study treatment with any agent(s) that have potential adverse drug-drug interactions (DDIs) with the study interventions; and
    * HCV disease has undergone appropriate work-up and is not advanced or associated with cirrhosis
17. Participants with untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of completed treatment at least 7 days prior to enrolment) are excluded. Participants with a false positive RPR (with negative treponemal test) or serofast RPR result (persistence of a reactive nontreponemal syphilis test despite history of adequate therapy and no evidence of re-exposure) may enroll after consultation with the Medical Monitor. Participants who completed treatment at least 7 days prior to enrolment are eligible.
18. Known or suspected presence of any major resistance mutations as defined by the international AIDS society (IAS)-United States of America (USA) resistance guidelines to DTG, 3TC, CAB or RPV in any resistance test result.
19. Participants with exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent (whichever is longer), prior to first dose of study treatment.
20. Participants with treatment with any of the following agents within 28 days of Screening:

    * radiation therapy
    * cytotoxic chemotherapeutic agents;
    * tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid, INH);
    * anti-coagulation agents, with the exception of the use of low dose acetylsalicylic acid (≤325 mg);
    * immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons. Note: Participants using short-term (e.g. ≤21 days) systemic corticosteroid treatment; topical, inhaled and intranasal corticosteroids are eligible for enrolment
21. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
22. Treatment with any agent with documented activity against HIV-1 in vitro within 28 days of first dose of study treatment. Treatment with acyclovir/valacyclovir is permitted.
23. Use of medications which are associated with Torsade de Pointes
24. Participants receiving any protocol-defined prohibited medication and who are unwilling or unable to switch to an alternate medication.
25. Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities.
26. Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the participant's participation in an interventional clinical trial.
27. Participant has estimated creatine clearance <30 milliliter per minute (mL/min) per 1.73 square meter (m^2) using the refitted, race-neutral Chronic Kidney Disease Epidemiology Collaboration (CKDEPIcr_R) method.
28. Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN); or ALT ≥3xULN and bilirubin ≥1.5xULN (with >35 percentage (%) direct bilirubin).
29. Participants known or suspected to have acquired HIV-1 concurrent with use of protease-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP) must be discussed with the Medical Monitor prior to enrolment.
30. Participant has a gluteal implant/enhancements (including fillers); or tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
31. Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study drugs.
32. Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
33. Participant is currently participating in, or anticipates being selected for, any other interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
[DTG/3TC]: Time to Virologic Suppression (HIV-1 Ribonucleic Acid [RNA] <50 Copies per Millilitre [c/mL]) From Baseline (Day 1) | Baseline (Day 1) up to Month 12
[CAB + RPV LA]: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL as per Snapshot Algorithm at Month 11 | Month 11

SECONDARY OUTCOMES:
[DTG/3TC]: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL as per Snapshot Algorithm at Month 12 | Month 12
[DTG/3TC]: Percentage of Participants With Plasma HIV-1 RNA Greater Than or Equal to (>=) 50 c/mL as Per Snapshot Algorithm | Month 12
[CAB + RPV LA]: Percentage of Participants With Plasma HIV-1 RNA >= 50 c/mL as Per Snapshot Algorithm | Month 11
Percentage of Participants With Plasma HIV-1 RNA <50 c/mL and <200 c/mL Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL and <200 c/mL Over Time | Up to and including Month 12
[CAB + RPV LA]: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL and <200 c/mL Over Time | Up to and including Month 11
Absolute Values for Plasma HIV-1 RNA (log10 c/mL) Through Day of choice | Up to and including Day of Choice (approximately 20 weeks)
Change From Baseline in Plasma HIV-1 RNA (log10 c/mL) Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Absolute Values for Plasma HIV-1 RNA (log10 c/mL) Through Month 12 | Up to and including Month 12
[DTG/3TC]: Change From Baseline in Plasma HIV-1 RNA (log10 c/mL) Through Month 12 | Baseline (Day 1) and up to and including Month 12
Absolute Values in Cluster of Differentiation 4 (CD4+) Cell Count Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
Change From Baseline in CD4+ Cell Count Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Absolute Values in CD4+ Cell Count Through Month 12 | Up to and including Month 12
[DTG/3TC]: Change From Baseline in CD4+ Cell Count Through Month 12 | Baseline (Day 1) and up to and including Month 12
[CAB + RPV LA]: Absolute Values of CD4+ Cell Count Through Month 11 | Up to and including Month 11
[CAB + RPV LA]: Change From Baseline in CD4+ Cell Count Through Month 11 | Baseline (Day 1) and up to and including Month 11
Percentage of Participants Meeting Confirmed Virologic Failure (CVF) Criteria Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Percentage of Participants Meeting CVF Criteria Over Time | Up to and including Month 12
[CAB + RPV LA]: Percentage of Participants Meeting CVF Criteria Over Time | Up to and including Month 11
Percentage of Participants With Disease Progression Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Percentage of Participants With Disease Progression Over Time | Up to and including Month 12
[CAB + RPV LA]: Percentage of Participants With Disease Progression Over Time | Up to and including Month 11
Percentage of Participants With Viral Resistance to CAB, RPV, DTG and 3TC Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
[DTG/3TC]: Percentage of Participants With Viral Resistance to CAB, RPV, DTG and 3TC Through Month 12 | Up to and including Month 12
[CAB + RPV LA]: Percentage of Participants With Viral Resistance to CAB, RPV, DTG and 3TC Through Month 11 | Up to and including Month 11
Percentage of Participants With Serious Adverse Events (SAEs), Drug Related Adverse Events (AEs) and AEs Leading to Discontinuation of Study Intervention Through Day of Choice | Up to and including Day of Choice (approximately 20 weeks)
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function which meets the definition of Hy's Law.
[DTG/3TC] Percentage of Participants With SAEs, Drug Related AEs and AEs Leading to Discontinuation of Study Intervention Over Time | Up to and including Month 12
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function.
[CAB + RPV LA] Percentage of Participants With SAEs, Drug Related AEs and AEs Leading to Discontinuation of Study Intervention Over Time | Up to and including Month 11
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function.
Change From Baseline in Total Treatment Satisfaction Score for HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) to Day of Choice | Baseline (Week 4) up to Day of Choice (approximately 20 weeks)
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied) producing a total score ranging from 0 to 66. Higher scores indicate a greater level of participant-reported satisfaction with their current therapy
Change From Baseline in Individual Item Score for HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) to Day of Choice | Baseline (Week 4) up to Day of Choice (approximately 20 weeks)
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied).
[DTG/3TC]: Change From Baseline in Total Treatment Satisfaction Score for HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Months 6 and 12 or up to Withdrawal | Baseline (Week 4) and at Month 6 and 12
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied) producing a total score ranging from 0 to 66. Higher scores indicate a greater level of participant-reported satisfaction with their current therapy
[DTG/3TC]: Change From Baseline in Individual Item Scores for HIVTSQs at Months 6 and 12 or up to Withdrawal | Baseline (Week 4) and at Month 6 and 12
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied).
[CAB + RPV LA]: Change From Baseline in Total Treatment Satisfaction Score for HIVTSQs at Months 5 and 11 or up to Withdrawal | Baseline (Week 4) and at Month 5 and 11
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied) producing a total score ranging from 0 to 66. Higher scores indicate a greater level of participant-reported satisfaction with their current therapy
[CAB + RPV LA]: Change From Baseline in Individual Item Scores for HIVTSQs at Months 5 and 11 or up to Withdrawal | Baseline (Week 4) and at Month 5 and 11
  HIVTSQ is a 12-item self-reported scale. Individual items are rated from 0 (very dissatisfied) to 6 (very satisfied).
Change From Baseline in Total Score of HIV Related Symptoms Assessed by Symptom Distress Module (SDM) Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
  SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 (complete absence of symptom) to 4 (very bothersome symptom). Overall score is calculated as the sum of the scores for each of the 20 items of the questionnaire and ranges from 0 (best health) to 80 (worst health).
Change From Baseline in Individual Bothersome Symptoms of HIV Assessed by SDM Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
  SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 (complete absence of symptom) to 4 (very bothersome symptom).
[DTG/3TC]: Change From Baseline in Total Score of HIV Related Symptoms Assessed by SDM at Month 6 and 12 | Baseline (Day 1) and at Month 6 and 12
  SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 (complete absence of symptom) to 4 (very bothersome symptom). Overall score is calculated as the sum of the scores for each of the 20 items of the questionnaire and ranges from 0 (best health) to 80 (worst health).
[DTG/3TC]: Change From Baseline in Individual Bothersome Symptoms of HIV Assessed by SDM at Month 6 and 12 | Baseline (Day 1) and at Month 6 and 12
  SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 (complete absence of symptom) to 4 (very bothersome symptom).
Change From Baseline in Health-Related Quality of Life Using World Health Organisation Quality of Life Brief version (WHOQoL-HIV-BREF) Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
  WHOQoL-HIV-BREF is a 31-item self-reported measure that addresses the 6 quality of life domains including (physical, psychological, level of independence, social relations, environment, spiritual) and 2 general health presence. The scales domain score ranges from 4 to 20. Higher scores indicate a better quality of life.
[CAB + RPV LA]: Change From Baseline in Health-Related Quality of Life Using WHOQoL-HIV-BREF at Month 5 and 11 | Baseline (Day 1) and at Month 5 and 11
  WHOQoL-HIV-BREF is a 31-item self-reported measure that addresses the 6 quality of life domains including (physical, psychological, level of independence, social relations, environment, spiritual) and 2 general health presence. The scales domain score ranges from 4 to 20. Higher scores indicate a better quality of life.
[DTG/3TC]: Change From Baseline in Health-Related Quality of Life Using WHOQoL-HIV-BREF at Month 6 and 12 | Baseline (Day 1) and at Month 6 and 12
  WHOQoL-HIV-BREF is a 31-item self-reported measure that addresses the 6 quality of life domains including (physical, psychological, level of independence, social relations, environment, spiritual) and 2 general health presence. The scales domain score ranges from 4 to 20. Higher scores indicate a better quality of life.
Change From Baseline in Anxiety and Depression Score Using Patient Health Questionnaire 9 (PHQ-9) Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
  PHQ-9 is a 9-item scale that assesses mood symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-27. Higher score indicates severe depression.
[DTG/3TC]: Change From Baseline in Anxiety and Depression Score Using PHQ-9 at Month 6 and 12 | Baseline (Day 1) and at Month 6 and 12
  PHQ-9 is a 9-item scale that assesses mood symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-27. Higher score indicates severe depression.
[CAB + RPV LA]: Change From Baseline in Anxiety and Depression Score Using PHQ-9 at Month 5 and 11 | Baseline (Day 1) and at Month 5 and 11
  PHQ-9 is a 9-item scale that assesses mood symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-27. Higher score indicates severe depression.
Change From Baseline in Anxiety and Depression Score Using General Anxiety Disorder 7 (GAD-7) Through Day of Choice | Baseline (Day 1) and up to and including Day of Choice (approximately 20 weeks)
  GAD-7 is a 7-item scale that assesses GAD symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-21. Higher score indicates severe anxiety.
[DTG/3TC]: Change From Baseline in Anxiety and Depression Score Using GAD-7 at Month 6 and 12 | Baseline (Day 1) and at Month 6 and 12
  GAD-7 is a 7-item scale that assesses GAD symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-21. Higher score indicates severe anxiety.
[CAB + RPV LA]: Change From Baseline in Anxiety and Depression Score Using GAD-7 at Month 5 and 11 | Baseline (Day 1) and at Month 5 and 11
  GAD-7 is a 7-item scale that assesses GAD symptoms over past two weeks. Each item is rated from 0 to 3 and yields a total score range of 0-21. Higher score indicates severe anxiety.
Percentage of Participants Providing Response to Single Item Bespoke Questions From Baseline to Day of Choice | Baseline (Day 1) and Day of Choice (approximately 20 weeks)
  Bespoke single-item questions are developed by ViiV Healthcare to assess concepts such as stigma, feelings about diagnosis, low mood/excitement relating to treatment.
[CAB + RPV LA]: Percentage of Participants Providing Response to Single Item Bespoke Questions From Day of Choice to Month 5 and 11 | Day of Choice (approximately 20 weeks) up to Month 5 and 11
  Bespoke single-item questions are developed by ViiV Healthcare to assess concepts such as stigma, feelings about diagnosis, low mood/excitement relating to treatment.
[DTG/3TC]: Percentage of Participants Providing Response to Single Item Bespoke Questions From Day of Choice to Month 6 and 12 | Day of Choice (approximately 20 weeks) up to Month 6 and 12
  Bespoke single-item questions are developed by ViiV Healthcare to assess concepts such as stigma, feelings about diagnosis, low mood/excitement relating to treatment.
[CAB + RPV LA]: Percentage of Participants Providing Response to Assessments Using ViiV Healthcare Developed Single Item Questionnaire From Day of Choice to Month 5 and 11 | Day of Choice (approximately 20 weeks) up to Month 5 and 11
  Bespoke single-item questions developed by ViiV Healthcare to assess long-acting specific concepts such as fear of disclosure of HIV status, adherence anxiety and daily reminder of HIV status.

CONTACTS AND LOCATIONS:
Locations (43):
- United States (15):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
- Argentina (4):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Rosario
- Canada (2):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (4):
  - GSK Investigational Site, La Cisterna
  - GSK Investigational Site, Providencia
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Temuco
- France (3):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Frankfurt am Main
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Italy (3):
  - GSK Investigational Site, Foggia
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
- GSK Investigational Site, Ponce, Puerto Rico
- Spain (7):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Granada
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/